CLINICAL TRIAL: NCT03634059
Title: A Study of Apatinib Plus EGFR-TKI as First Line Treatment in Patients With Non-squamous NSCLC Harboring EGFR Mutations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, LiuJunFeng, Principal Investigator, Hebei Medical University Fourth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRA-L01
Record Dates: First submitted 2018-07-12; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: NSCLC
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib (Experimental): apatinib 500mg qd po plus Erlotinib 150mg qd po / apatinib 500mg qd po plus Icotinib 125mg tid po
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — apatinib 500mg qd po plus Erlotinib 150mg qd po / apatinib 500mg qd po plus Icotinib 125mg tid po

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of apatinib plus EGFR-TKI as first line treatment in patients with non-squamous NSCLC harboring EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 to 75 years old (man or female);
2. Pathologically diagnosed with non-squamous NSCLC;
3. Imageology diagnosed with locally advanced/metastatic or recurrent (stage ⅢB - IV);
4. Histologically or cytologic confirmed，harboring an activating EGFR mutation (19del or 21 L858R);
5. None previous chemotherapy or targeted therapy.（NOTE: neoadjuvant and adjuvant therapy is allowed）;
6. At least one measurable lesion (measuring≥10mm on spiral CT scan, satisfying the criteria in RECIST1.1)；
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
8. Major organ function has to meet the following criteria:

   1. HB≥90g/L；
   2. ANC≥1.5×109/L；
   3. PLT≥80×109/L；
   4. ALT and AST≤2.5ULN, but≤5ULN if the transferanse elevation is due to liver metastases;
   5. TBIL≤1.5ULN;
   6. Serum creatinine≤1.25ULN; Endogenous creatinine clearance rate>45 ml/min;
9. Life expectancy greater than or equal to 3 months;
10. Women of childbearing age must have contraceptive measures or have test pregnancy (serum or urine) enroll the study before 7 days, and the results must be negative, and take the methods of contraception during the test and the last to have drugs after 8 weeks. Men must be contraception or has sterilization surgery during the test and the last to have drugs after 8 weeks;
11. Participants were willing to join in this study, and written informed consent, good adherence, cooperate with the follow-up.

Exclusion Criteria:

1. Have high blood pressure and antihypertensive drug treatment can not control (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
2. Patients who suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female ≥ 470 ms). Grade III-IV cardiac insufficiency according to New York Heart Association(NYHA) criteria or echocardiography check: left ventricular ejection fraction (LVEF)<50%;
3. Radiologically documented evidence of major blood vessel invasion or encasement by cancer;
4. A variety of factors influencing oral drugs (such as unable to swallow, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc);
5. Patients with tendency of gastrointestinal bleeding, including the following: a local active ulcerative lesions, and defecate occult blood (++). Has melena and hematemesis in two months;
6. Coagulant function abnormality (INR > 1.5 ULN, APTT > 1.5 ULN), with bleeding tendency;
7. Patients with pregnant or planning a pregnancy;
8. Patients with other malignant tumors within 5 years (except for the treated skin basal cell carcinoma and cervical carcinoma in situ);
9. History of psychiatric drugs abuse and can't quit or patients with mental disorders;
10. Less than 4 weeks from the last clinical trial;
11. The researchers think inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2019-08-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | evaluated in two years since the treatment began
  Baseline to measured date of progression or death from any cause

SECONDARY OUTCOMES:
Objective response rate | tumor assessment every 8 weeks，up to two years
  Baseline to measured stable disease
Disease control rate (DCR) | tumor assessment every 8 weeks，up to two years
  Baseline to measured progressive disease
Overall survival (OS) | the first day of treatment to death or last survival confirm date，up to two years
  Baseline to measured date of death from any cause
Adverse events | evaluated in the two years since the treatment began according to the Common Terminology Criteria for Adverse Events Version 4.0
  throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Junfeng Liu, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Junfeng Liu, Shijiazhuang, Hebei, China